## Institutional Review Board Consent to Participate in Research

Principal Investigator: Britany Raymond Version Date: 10/18/2020

Study Title: Perioperative Ketamine Infusion and Inpatient Opioid Consumption

Institution/Hospital: Vanderbilt University Medical Center

## SHORT FORM WRITTEN INFORMED CONSENT DOCUMENT

This document must be written in a language <u>understandable</u> to the subject and should be attached to a written summary of the information that is presented orally.

You are being asked to take part in a research study.

Before you agree, the study doctor must tell you about:

- (i) the reason for doing the study, the things that will be done and how long you will be in the study;
- (ii) any tests or treatments that are experimental;
- (iii) any risks or side effects you can expect, and good effects that might come from the study;
- (iv) other treatments you could get if you decide not to be in the study; and

When any of the following things apply, the study doctor must also tell you about:

- (i) the possibility of other risks that are not known;
- (ii) reasons why the study doctor may take you out of the study;
- (iii) what will happen if you decide to stop being in the study;

A description of this clinical trial will be available on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

If you have any questions about this research study or if you feel you have been hurt because of this study, please feel free to contact Britany L. Raymond, MD at 615-322-8476

You can also contact my Faculty Advisor, Matthew D. McEvoy at 615-936-5194.

If you cannot reach the research staff, please page the study doctor at 615-936-5194.

For additional information about giving consent or your rights as a participant in this study, contact the Institutional Review Board Office at (615) 322-2918 or toll free at (866) 224-8273.

You do not have to be in this research study. You may choose not to be in this study and get other treatments without changing your healthcare, services or other rights. You can stop being in this study at any time.

## STATEMENT BY PERSON AGREEING TO BE IN THIS STUDY The research study has been explained to me verbally. All my questions have been answered, and I freely and voluntarily choose to take part in this study. Signature of Participant Date Date

**Institutional Review Board** 

**VANDERBILT** 

06/01/2017